CLINICAL TRIAL: NCT03320915
Title: Efficacy and Safety of High Dose Vitamin D Supplementation in Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Efficacy and Safety of High Dose Vitamin D Supplementation in Patients Undergoing HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University (Other)
Responsible Party: Principal Investigator, Youngil Koh, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1702-040-830
Record Dates: First submitted 2017-10-22; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cholecalciferol (Experimental): Cholecalciferol 5mg (200,000 IU)
  Interventions: Drug: Cholecalciferol
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Drug: Cholecalciferol — Cholecalciferol 5mg (200,000 IU) up to maximum of three times during 1 year follow-up period according to measured 25(OH)D3 level.
  Other Names: Caldiferol
  Arms: Cholecalciferol

SUMMARY:
Graft-versus-host-disease (GVHD) is common complication of hematopoietic stem cell transplantation. Vitamin D deficiency has been shown to be associated with increased risk of chronic GVHD in previous clinical studies. The purpose of this research is to investigate the effect of vitamin D supplementation in patients undergoing hematopoietic stem cell transplantation

DETAILED DESCRIPTION:
Hematopoietic stem cell transplant candidates are randomized to vitamin D supplementation or usual care. Five milligrams (200,000 IU) of cholecalciferol is injected to intervention group before stem cell transplantation. Additional supplementation of cholecalciferol during follow-up period is determined according to the level of 25(OH)D3. The primary outcome is the incidence of chronic GVHD which is determined according to IBMTR criteria. The secondary outcome consists of the incidence of acute GVHD, incidence and severity of vitamin D deficiency, and serum concentration of 25(OH)D3. Study investigators expect that supplementation of vitamin D may improve the outcome of stem cell transplantation by reducing the incidence of chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Adults with ≥ 18 years old
* Diagnosed with hematologic maligancies
* Planned to undergo allogeneic stem cell transplantation

Exclusion Criteria:

* Hypercalcemia (ionized serum calcium level [iCa] > 1.3 mmol/L, corrected serum calcium level > 10.5 mg/dL)
* Impaired renal function (Serum creatinine ≥ 2.4 mg/dL)
* Not in complete remssion (except for myelodysplastic syndrome and myeloproliferative neoplasm)
* Consent withdrawal
* Considered inadequate under investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Chronic GVHD | Up to 1 year
  Events will be graded according to IBMTR criteria

SECONDARY OUTCOMES:
Acute GVHD | Up to 100 days
  Events will be graded according to IBMTR criteria
Vitamin D deficiency | Up to 1 year
  Severity and incidence of Vitamin D deficiency
25(OH)D3 | Up to 1 year
  Serum concentration of 25(OH)D3

CONTACTS AND LOCATIONS:
Overall Officials: Youngil Koh, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea